CLINICAL TRIAL: NCT04625478
Title: Clinical Relevance of Intracellular Staphylococci in BOne and Joint Infections
Acronym: CRISBO
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 229
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Bone and Joint Infection; Staphylococcus
Keywords: Bone and Joint Infection; Staphylococcus; intracellulare

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients having had an osteo-articular infection with Stahylococcus: Patients having had an osteo-articular infection with Stahylococcus managed at the Croix Rousse hospital
  Interventions: Other: Patients having had an osteo-articular infection with Stahylococcus

INTERVENTIONS:
Other: Patients having had an osteo-articular infection with Stahylococcus — Immunostaining targeting staphylococci and components will be performed on tissue samples collected from patients with osteo-articular infection

SUMMARY:
Different mechanisms have been proposed to explain the pathophysiology of chronic staphylococcal BJI, including biofilm formation and the ability of staphylococci to be internalized and to survive within cells. The intracellular localization of staphylococci is well documented by in vitro studies, however, few studies have shown the presence of intracellular staphylococci in clinical specimens from patients with BJI.

The aim of the CRISBO study is to document the clinical relevance of intracellular staphylococci in the context of BJI. Immunostaining targeting staphylococci and components will be carried out on tissue samples taken from patients with BJI during their treatment (samples similar to those used for routine diagnosis in pathology). Our objectives are to identify whether intracellular staphylococci are observable in these samples and if so, in which cell type (s) are they housed.

ELIGIBILITY:
Inclusion Criteria:

* patients having had an osteo-articular infection with Staphylococci

Exclusion Criteria:

-

Ages: 18 Years to 95 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients having had an osteo-articular infection with Staphylococci managed at the Croix-Rousse Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
detection of intracellular staphylococci | 2 months
  to explore if intracellular staphylococci can be observed on samples of patient having an osteo-articular infection with staphylococci
rate of localisation of intracellular staphylococci | 2 months
  to explore where in what type of celles they can be observed on samples of patient having an osteo-articular infection with staphylococci

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/